CLINICAL TRIAL: NCT07324408
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Multiply Ascending Dose of NH102 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study of NH102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH102-12
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NH102 3mg (Experimental): NH102 3mg or NH102 placebo-matching, tablet, orally, bid (at approximately 8:00 AM and 8:00 PM). The morning doses on D1 and D7 (around 8:00 AM) are to be given under fasting conditions. A total of 13 consecutive doses are administered. For fasting doses: fast for at least 10 hours before dosing, fast for 4 hours after dosing, and no water intake 1 hour before and 1 hour after dosing.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 10mg (Experimental): NH102 10mg or NH102 placebo-matching, tablet, orally, bid (at approximately 8:00 AM and 8:00 PM). The morning doses on D1 and D7 (around 8:00 AM) are to be given under fasting conditions. A total of 13 consecutive doses are administered. For fasting doses: fast for at least 10 hours before dosing, fast for 4 hours after dosing, and no water intake 1 hour before and 1 hour after dosing.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 15mg (6 mg→10 mg→15 mg） (Experimental): NH102 6/10/15 mg or NH102 placebo-matching, tablet, orally, bid (at approximately 8:00 AM and 8:00 PM). Days 1-2: 6 mg, bid; Days 3-5: 10 mg, bid; Days 6-9: 15 mg, bid (administered only once on Day 9), for a total of 17 consecutive doses. The morning doses on D1 and D9 (around 8:00 AM) are to be given under fasting conditions. For fasting doses: fast for at least 10 hours before dosing, fast for 4 hours after dosing, and no water intake 1 hour before and 1 hour after dosing.
  Interventions: Drug: NH102; Drug: Placebo
- NH102 20mg (10 mg→15 mg→20 mg） (Experimental): NH102 10/15/20 mg or NH102 placebo-matching, tablet, orally, bid (at approximately 8:00 AM and 8:00 PM). Days 1-2: 10 mg, bid; Days 3-5: 15 mg, bid; Days 6-9: 20 mg, bid (administered only once on Day 9), for a total of 17 consecutive doses. The morning doses on D1 and D9 (around 8:00 AM) are to be given under fasting conditions. For fasting doses: fast for at least 10 hours before dosing, fast for 4 hours after dosing, and no water intake 1 hour before and 1 hour after dosing.
  Interventions: Drug: NH102; Drug: Placebo

INTERVENTIONS:
Drug: NH102 — tables orally
Drug: Placebo — tables orally

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of NH102 when administered as multiple oral dose at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called NH102. NH102 is being tested to treat people who have depression. This study will look at the safety, tolerability and PK of NH102 in healthy participants.

The study may enroll up to 30-40 participants. Participants will be randomly assigned within each cohort to receive NH102 or placebo which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need). The study consists of four dose groups: 3 mg (fixed dose), 10 mg (fixed dose), 15 mg (starting at 6 mg, then escalated to 10 mg, and finally to 15 mg), and 20 mg (starting at 10 mg, then escalated to 15 mg, and finally to 20 mg). Each group enrolls 10 subjects, with 8 receiving NH102 and 2 receiving placebo. For the third and fourth dose groups (15 mg and 20 mg) that follow a titration dosing regimen, each includes 2 sentinel subjects (both male). The two sentinel subjects may be dosed simultaneously. Only after both sentinel subjects complete all 17 doses (with a single dose administered on Day 9) and are observed for at least 24 hours, along with preliminary confirmation of safety, may the remaining subjects in the same dose group proceed with dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 (both inclusive) years old when signing the informed consent.
2. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18.5 and ≤28 kg/m2 at screening.
3. Subjects voluntarily participate and sign the informed consent after understanding the purpose, content, procedures and possible risks of the trial.
4. The subjects will be able to communicate well with the investigators, be willing and able to comply with the lifestyle restrictions specified in the protocol, and cooperate to complete the study.

Exclusion Criteria:

1. The investigator determined that the subjects' present medical history and past medical history had any disease or dysfunction that would affect the clinical trial, including but not limited to diseases of the central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, hematological system, etc.
2. There is any surgical condition or disease that may significantly affect the absorption, distribution, metabolism and excretion of drugs, or may harm to the subjects participating in the trial; such as history of gastrointestinal operations (gastrectomy, gastroenterostomy, enterectomy, etc.), urinary tract obstruction or dysuria, gastroenteritis, digestive tract ulcers, history of gastrointestinal bleeding, etc.
3. Subjects with past history of allergy to drugs or allergic disease.
4. Subjects with currently or past history of mental disorders and brain functional disorders.
5. According to the Columbia suicide severity scale (C-SSRS), subjects were at risk of suicide or were at risk of suicide based on the clinical judgment of the researchers, or with past history of self-injurious behavior.
6. Subjects have history of drug abuse or positive urine drug tests at screening within 1 year prior.
7. Subjects have history of alcohol abuse(i.e.,criteria are per week consumption more than 14 standard units(1 unit =360mL beer or 45mL 40% alcohol of Chinese liquor or 150mL wine)or positive alcohol breath tests at screening within 1 year prior.
8. Average amount of daily smoking>5 cigarettes at screening 3 months prior.
9. Those who have special requirements for food, cannot follow a uniform diet or have difficulty swallowing.
10. Female subjects who are pregnant and lactating ; and those who refuse to use effective non-drug contraceptive measures (such as abstinence, intrauterine device) or have planned to donate sperm or ovum throughout the study period and within 3 months after the end of the study.
11. Abnormal vital signs, lab and ECG indicators, as determined by the researcher, and clinically significant (e.g., male QTC > 450ms female > 470ms,corrected by Friericia ).
12. Subjects who resting heart rate <55 beats/min or >100 beats/min; systolic blood pressure <90mmHg or >140mmHg; diastolic blood pressure <60mmHg or >90mmHg.
13. Subjects who hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab), or HIV antibody (HIV-Ab), or syphilis serum reaction (TRUST) is non-negative.
14. Subjects who participated in any clinical trial within 3 months before medication.
15. Subjects have history of blood donations of 400 mL within 3 months before enrollment; 200 mL within 1 month before enrollment; or have history of using blood products.
16. Subjects who had a history of surgery within 3 months prior to enrollment, or did not recover from surgery, or had an expected surgical plan during the study period.
17. Subjects who had taken any drugs, including prescription and over-the-counter drugs within 2 weeks prior to enrollment.
18. Subjects who directly related to this clinical trial.
19. Subjects have poor compliance or other problems that the researchers believe that it is not suitable for participating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)
Number of participants with change in laboratory parameters following treatment administration | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)
  The laboratory parameters include hematology, clinical chemistry, coagulation and urinalysis.
Number of participants with change in vital sign measurements following treatment adminstration | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)
  The items of vital sign include blood pressure, heart rate, body temperature and respiratory rate.
Number of participants with change in physical examination following treatment administration | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)
Number of participants with change in 12-lead ECG following treatment administration | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)
Number of participants with change in Columbia-suicide severity rating scale (C-SSRS) score | Baseline up to Day 9 ( the 3 mg and 10mg dose groups) or Day 10 (the 15 mg and 20 mg dose groups)

SECONDARY OUTCOMES:
Plasma PK parameters-Maximum plasma concentration (Cmax) after single-dose administration | From pre-dose to 12 hours (before the second administration on Day 1)
Plasma PK Parameters-Time for maximum plasma concentration (Tmax) | From pre-dose to 12 hours (before the second administration on Day 1), and from pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Area Under Curve from zero to 24 hours (AUC0-12h) | From pre-dose to 12 hours (before the second administration on Day 1)
Plasma PK Parameters-Maximum observed drug concentration at steady state (Cmax,ss) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Minimum observed drug concentration at steady state (Cmin,ss) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK-Parameters-Average drug concentration at steady state (Cav,ss) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Area Under Curve from time zero to the last time point with a measurable concentration (AUC0-t) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Area Under Curve from zero to infinity (AUC0-∞) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Area Under Curve over a dosing interval at steady state (AUCss) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Apparent total body clearance at steady state after extravascular administration (CLss/F) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Trough drug concentration (Ctrough) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Degree of Fluctuation (DF) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Terminal elimination rate constant (λz) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Relative bioavailability based on AUC [Ra(AUC)] | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Terminal half-life (t1/2z) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.
Plasma PK Parameters-Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | From pre-dose on Day 7 to 48 hours (Day 9) for the 3 mg and 10 mg dose groups, or from pre-dose on Day 9 to 24 hours (Day 10) for the 15 mg and 20 mg dose groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No